CLINICAL TRIAL: NCT02062450
Title: Multicentre, Observational Study Evaluating the Clinical and Radiological Outcomes of Hip Arthroplasty Using the Dual Mobility Cup
Brief Title: Observational Study Evaluating Outcomes of Hip Arthroplasty Using Tornier Dual Mobility Acetabular Cup
Status: Completed | Type: Observational
Sponsor: Stryker Trauma and Extremities (Industry)
Responsible Party: Sponsor
Other Study IDs: 1204-T-DOUBLEMOB-RM
Record Dates: First submitted 2014-02-11; First posted 2014-02-13 (Estimated); Results first posted 2016-05-16 (Estimated); Last update posted 2017-05-04 (Actual); Status verified 2017-05

CONDITIONS: Primary Osteoarthritis; Post-traumatic Osteoarthritis of Hip Nos; Femur Head Necrosis; Femur Neck Fracture; Congenital Dislocations
Keywords: Arthroplasty; Hip Replacement; Acetabular cup; Dual mobility; Hip revision surgery
MeSH Terms: conditions — Femur Head Necrosis; Femoral Neck Fractures | interventions — Reoperation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Primary surgery with Dual Mobility Cup: Patients having a Primary Hip acetabular replacement, using a Dual Mobility Cup.
  Interventions: Device: Primary surgery with Dual Mobility Cup
- Revision surgery with Dual Mobility Cup: Patients having a Revision Hip acetabular replacement, using a Dual Mobility Cup.
  Interventions: Device: Revision surgery with Dual Mobility Cup

INTERVENTIONS:
Device: Primary surgery with Dual Mobility Cup — Hip joint replacement with a hip prosthesis including a Dual Mobility cup to replace the acetabular component.
  Groups: Primary surgery with Dual Mobility Cup
Device: Revision surgery with Dual Mobility Cup — Hip joint replacement with a hip prosthesis including a Dual Mobility cup to replace the acetabular component.
  Groups: Revision surgery with Dual Mobility Cup

SUMMARY:
The purpose of this study is to demonstrate the performance and reliability of Tornier "Dual Mobility Cup" used during primary total hip replacement or hip replacement revision surgery at least 24 months post-insertion.

DETAILED DESCRIPTION:
The PURPOSE of this study is to demonstrate the performance and reliability of the Tornier "Dual Mobility Cup" used during primary total hip replacement or hip replacement revision surgery at a minimum of 24 months post-implantation. The primary endpoint is to determine the dislocation rate observed during post-surgical follow-up. The secondary endpoints are to assess, in the short-term, the following: clinical performance on the basis of clinical scores and hip mobility; radiological performance, particularly in terms of positioning and fixation of the implant; as well as the reliability of the implantation of this acetabular cup on the basis of any complications observed

ELIGIBILITY:
Inclusion Criteria:

* men and women aged over 18, undergoing total hip replacement with insertion of a Dual Mobility acetabular cup between October 2010 and October 2011,
* capable of attending the 2-year follow-up visit;
* capable of understanding the information about the study and agreeing to take part in it.

Exclusion Criteria:

* patients with tumoral pathology.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The global cohort: All the patients who received a Tornier Dual Mobility acetabular cup between October 2010 and October 2011 and who we were able to be contacted by phone.
  "Primary replacement" group: All the patients who received a Tornier Dual Mobility acetabular cup between October 2010 and October 2011 for primary hip replacement and who were seen for their follow-up visit at 2 years post-procedure.
  "Revision" group: All patients who received a Tornier Dual Mobility acetabular cup between October 2010 and October 2011 for revision surgery and who were seen for their follow-up visit at 2 years post-procedure.
  All the performance criteria were analysed for the patients in the "Primary replacement" and "Revision" groups
Sampling Method: Probability Sample
Enrollment: 379 (Actual)
Dates: Start 2013-05; Primary Completion 2013-11 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christophe Hulet, MD, PR, Principal Investigator — Caen University Hospital, FR

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 472 patients who underwent hip arthroplasty with a Dual Mobility Cup between September 2010 and December 2011, in the 5 participating centers, have been identified.
  379 out of them have been successfully reached by phone to be convoked for their 2-year postoperative follow-up visit. The other 93 patients were considered "lost to follow-up".
Pre-assignment Details: Of the 379 contacted patients, 255 came to visit their surgeons for the 2-year follow-up. The other 124 who declined to visit were evaluated by phone for safety criteria.
Groups:
- Hip Acetabular Replacement, Using a Dual Mobility Cup.: Studied cohort includes 2 subgroups :
  * Patients with primary hip replacement.
  * Patients with revision surgery.
Period: Overall Study
Arm/Group | Hip Acetabular Replacement, Using a Dual Mobility Cup.
Started | 379 (379 patients were successfully reached by phone and convoked for the 2-year follow-up visit.)
Per Protocol Cohort | 255 (255 patients attended their 2-year follow-up visit.)
Completed | 255
Not Completed | 124
Not completed — No follow-up visit | 124

BASELINE CHARACTERISTICS:
Population: A total of 255 patients were included in the Global Study Cohort of which 191 had a Primary Hip surgery and 64 had a Revision Hip surgery.
Groups:
- Primary Surgery: Patients who underwent a primary hip replacement surgery with Dual Mobility Cup
- Revision Surgery: Patients who underwent a revision hip replacement surgery with Dual Mobility Cup
- Total: Total of all reporting groups
Arm/Group | Primary Surgery | Revision Surgery | Total
Number analyzed (Participants) | 191 | 64 | 255
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.7 (9.4) | 71.3 (11.5) | 72.2 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 87 | 33 | 120
  Male | 104 | 31 | 135
Region of Enrollment [Number; unit: participants]
  France | 191 | 64 | 255

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With an Implant Dislocation After Surgery
Description: The primary safety outcome (implant dislocation) was assessed by a single question to the patients : Did you experience any implant dislocation since your surgery ? Positive answers were quantified.
Time Frame: 2-year postoperative
Population: 2 implants dislocations were reported in the 379 patients making up the Total Safety Population, of which 1 concerned a Primary surgery and the other concerned a Revision surgery. In both cases, orthopaedic reduction was performed without changing the implant.
Measure: Number; unit: participants
Groups:
- Total Safety Population: All patients implanted between Sept 2010 and Dec 2011 who were reached by phone and could answer to the safety questions.
Arm/Group | Total Safety Population
Number analyzed (Participants) | 379
participants | 2

2. Primary Outcome: Percentage of Participants With an Implant Dislocation After Surgery (= Dislocation Rate)
Description: as for outcome 1
Time Frame: 2-year postoperative
Measure: Number; unit: percentage of participants
Arm/Group | Total Safety Population
Number analyzed (Participants) | 379
percentage of participants | 0.53

3. Secondary Outcome: Clinical Performance - PMA Score
Description: Postel-Merle-d'Aubigné (PMA) score is known since 1954 and is a very widespread mean of evaluating the clinical function of the hip by the physician.
  It contains three items: pain, function and hip mobility, each noted on 6 points (0 is the worst possible score and 18 is the best possible score) :
  * a score between 15 and 18 points is defined as good,
  * a score between 12 and 14 points is defined as average,
  * a score inferior to 12 is defined as bad
Time Frame: 2 years postoperative
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Primary Surgery Sub-group: Patients who undergone a primary hip replacement surgery
- Revision Sub-group: patients who undergone a revision hip replacement surgery
Arm/Group | Primary Surgery Sub-group | Revision Sub-group
Number analyzed (Participants) | 191 | 64
units on a scale
  Baseline | 10.8 (2.6) | 9.3 (3.3)
  2-y FU visit | 16.4 (2.5) | 15.2 (2.6)
  Improvement at 2-y FU vs Baseline | 6.1 (2.6) | 5.9 (3.8)

4. Secondary Outcome: Clinical Performance - HOOS Score
Description: The HOOS (Hip disability and Osteoarthritis Outcome Score) is a patient questionnaire evaluating patients' feelings about their operated hip. It consists of 40 questions divided into 5 subgroups: pain, symptoms, daily living, quality of life, sports and recreational activities. Each category is scored on 100 points, 0 being the worse outcome and 100 the best outcome.
Time Frame: 2 years postoperative
Measure: Mean (Standard Deviation); unit: units on a scale of 100
Arm/Group | Primary Surgery Sub-group | Revision Sub-group
Number analyzed (Participants) | 191 | 64
units on a scale of 100
  Pain | 91.8 (13.6) | 86.4 (15.1)
  Symptoms | 87.5 (15.1) | 84.5 (13.4)
  Daily living | 84.2 (22.0) | 76.6 (18.2)
  Sports and recreational activities) | 63.8 (33.2) | 43.2 (27.6)
  Quality of Life | 85.2 (20.5) | 67.0 (26.7)

5. Secondary Outcome: Clinical Performance - HARRIS Score
Description: The HARRIS score is a physician questionnaire assessing hip pain, function and mobility on a total of 100 points, 100 being the maximum score. A result between 90 and 100 points is considered "excellent", between 80 and 90 "good", between 70 and 80 "mediocre" and less than 70 "poor".
Time Frame: 2-year postoperative
Measure: Number; unit: percentage of partipants
Arm/Group | Primary Surgery Sub-group | Revision Sub-group
Number analyzed (Participants) | 191 | 64
percentage of partipants
  Excellent | 64 | 40
  Good | 13 | 16
  Mediocre | 10 | 19
  Poor | 12 | 24

6. Primary Outcome: Implant Survivorship
Description: Implant survivorship criteria was assessed by investigators during patients visits : is the implanted device still in place 2 years after surgery ? Negative answers were quantified.
Time Frame: 2-year postoperative
Measure: Number; unit: percentage of implants
Arm/Group | Total Safety Population
Number analyzed (Participants) | 379
percentage of implants | 99.5

ADVERSE EVENTS:
Time Frame: 2 years postoperative
Groups:
- Primary Surgery Sub-group: Patients who underwent a Primary Hip Replacement surgery
- Revision Surgery Sub-group: Patients who underwent a Revision Hip Replacement surgery
Arm/Group | Total Safety Population | Primary Surgery Sub-group | Revision Surgery Sub-group
Serious Adverse Events (participants affected / at risk) | 11/379 | 2/191 | 3/64
Other Adverse Events (participants affected / at risk) | 11/379 | 4/191 | 2/64
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Total Safety Population (N=379) | Primary Surgery Sub-group (N=191) | Revision Surgery Sub-group (N=64)
Dual Mobility Cup dislocation (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 0 (0) — Orthopedic reduction only - No Revision surgery
Revision surgery for Implant Mobilisation (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Revision surgery for Implant Loosening (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Revision surgery for Infection (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1) | 1 (1)
Revision surgery for Implant Malposition (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Revision surgery for Instability (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Transfemoral Amputation (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Osteosynthesis surgery (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Osteolysis surgery (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Total Safety Population (N=379) | Primary Surgery Sub-group (N=191) | Revision Surgery Sub-group (N=64)
Infection without revision surgery (Musculoskeletal and connective tissue disorders) | 4 (4) | 1 (1) | 1 (1)
Recurrent Pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 3 (3) | 0 (0)
Wound affection (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0) | 0 (0)
Asymptomatic implant mobilisation (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less